CLINICAL TRIAL: NCT00565526
Title: Clinical and Laboratory Evaluation of the Autonomic Nervous System in Primary Sjogren's Syndrome
Brief Title: Evaluation of the Role of the Autonomic Nervous System in Sj(SqrRoot)(Delta)Gren s Syndrome
Status: Completed | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080018; 08-D-0018
Record Dates: First submitted 2007-11-29; First posted 2007-11-30 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2014-04-10

CONDITIONS: Sjogren's Syndrome; Dysautonomia
Keywords: Autonomic Nervous System; Sjogren's Syndrome; Pathogenesis; Cholinergic; Parasympathetic; Sjogren Syndrome
MeSH Terms: conditions — Sjogren's Syndrome; Autonomic Nervous System Diseases

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

Sj(SqrRoot)(Delta)gren s Syndrome (SS) is an autoimmune disease that affects the glands that produce saliva and tears, causing dry eyes and dry mouth.

Researchers do not know the exact cause of SS, but they believe that it may be caused by abnormalities in the autonomic nervous system (ANS) that stimulate these glands.

Objectives:

To better understand ANS function in patients with SS.

To compare information about ANS function in healthy individuals and in patients with SS.

Eligibility:

Patients with Sj(SqrRoot)(Delta)gren s Syndrome who are 18 years of age and older, and who are not pregnant or breastfeeding.

Participants will be asked to taper or discontinue the use of certain medications or dietary supplements before the ANS testing.

Participants must be willing to discontinue the use of alcohol and tobacco 24 hours prior to testing.

Design:

The study will require one inpatient admission and/or outpatient visits to the NIH Clinical Center.

The following tests and procedures will be performed:

* Saliva, tear, and sweat production measurements to evaluate the function of glands.
* Testing of changes to the cardiovascular system, including blood pressure and blood flow testing, and an electrocardiogram designed to evaluate hemodynamic changes controlled by the ANS.
* Testing of changes to the gastrointestinal system, including a swallowing assessment study, barium swallow study, and gastric emptying study designed to evaluate gastrointestinal function controlled by the ANS.
* Tests to evaluate the ANS function in response to certain drugs (edrophonium, glucagon and acetylcholine).
* Self-reported questionnaire on ANS function and emotional/psychological well-being.

Additional procedures and tests may include the following:

* Blood samples.
* Optional skin biopsy to study sweat glands and nerve supply of the skin.

DETAILED DESCRIPTION:
Sj(SqrRoot)(Delta)gren s syndrome (SjS) is a systemic exocrinopathy that affects as high as 5 percent of the population. It is manifested predominantly as dry eyes, dry mouth, and fatigue. The exocrinopathy can be encountered alone (primary SjS) in approximately one half of the patients or in the presence of another autoimmune disorder such as rheumatoid arthritis, systemic lupus erythematosus, or systemic sclerosis (secondary SjS). The most widely accepted classification for SjS is the American-European consensus classification criteria for SjS.(Vitali, Bombardieri et al. 2002)

Current understanding about the pathogenesis of SjS stems from the assumption that the autoimmune destruction of the exocrine glands leads to their hypofunction and symptoms of dryness. The existing evidence however does not fully support this assumption and cannot explain the underlying pathogenic mechanisms of SjS for the following reasons: 1) Discordance between severely affected function and abundance of histologically normal and ex vivo functional salivary glands; 2) at least 20% of patients have no evidence of systemic autoimmunity; 3) Animal models of SjS develop glandular dysfunction long before they develop autoimmunity; 4) Dryness and related symptoms respond poorly to immunosuppressive, including newer biologics, but fairly well to secretagogues such as pilocarpine. 5) No pathogenic antibodies or target epitopes have been identified to date to unify the pathogenesis of the syndrome.

All exocrine glands are innervated by the autonomic nervous system (ANS) and dysautonomia can mimic the phenotype of SjS, particularly cardinal manifestations, such as xerostomia and xerophthalmia. Thus we hypothesize that ANS dysfunction is central to the pathogenesis of SjS and propose to systematically study the ANS function in our cohort of patients with primary SjS compared with normative data from age and sex-matched controls. This protocol calls for a comprehensive evaluation of autonomic function, using physiological, neuropharmacologic, neurochemical, and imaging approaches, to identify consistent distinctive patterns of ANS involvement in SjS and thereby improve the diagnosis and understanding of pathophysiologic mechanisms of SjS.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Diagnosis of primary Sjogren s syndrome based on American-European Consensus Group Sjogren s syndrome classification criteria or healthy volunteers.
  2. Both genders and all minorities.
  3. Age at entry at least 18 and less than 65 years.

EXCLUSION CRITERIA:

1. Current use of medications known to significantly influence the activity of the sympathetic or parasympathetic nervous system if they cannot be held safely at the time of ANS testing
2. Known co-existing diagnosis of ANS dysfunction (for healthy volunteers)
3. Medications-requiring diabetes mellitus
4. Diabetic autonomic neuropathy
5. Vitamin B12, folate deficiency, requiring replacement
6. Hepatic failure (AST or ALT greater than 1.5 x upper limit of normal)
7. Renal failure (GFR less than 30 ml/min, as estimated by the MDRD)
8. Congestive heart failure (Class II-IV)
9. Refractory ventricular arrhythmias
10. Symptomatic coronary heart disease
11. Previously established diagnosis of sinus node dysfunction
12. Severe anemia (Hgb less than 8)
13. Psychosis
14. Pregnant or lactating women
15. A candidate subject is excluded if, in the judgment of the Principal Investigator, protocol participation would place the subject at substantially increased acute medical risk.
16. Not able to provide informed consent

Medications: A candidate subject is excluded if clinical considerations require that the subject continue treatment with a drug likely to interfere with the scientific results i.e. a tricyclic antidepressant or fludrocortisone. Subjects with known or suspected allergy or hypersensitivity to any test drug are excluded from receiving that drug. Subjects who must take medications daily in the following categories are excluded: tricyclic antidepressants, beta blockers, barbiturates, if they cannot be safely held during testing. Subjects unable to discontinue nicotine or alcohol temporarily are excluded. Subjects are not to discontinue any medications before the subject or the subject s physician discusses this with the Principal Investigator, Dr. Nikolov, or the Associate Investigator, Dr. Goldstein. If it is decided that discontinuing medications would be unsafe, then the subject is excluded from the study. Subjects must discontinue use of alcohol and tobacco throughout the period of testing in the protocol.

Herbal Medicines and Dietary Supplements: Certain herbal medicines or dietary supplements are known or suspected to interfere with the experimental results, and such herbal medicines or dietary supplements must be discontinued before enrollment in the study. For many herbal medicines or dietary supplements, the mechanisms of action and therefore the possible effects on the experimental results are unknown. In cases where the subjects wish to continue their herbal medicines or dietary supplements while on study, and search of the available medical literature fails to identify effects that are known or expected to interfere with the experimental results, then the subjects may participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-11-26; Study Completion 2014-04-10

CONTACTS AND LOCATIONS:
Overall Officials: Stamatina J Danielides, M.D., Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Sharma RV, Mathur SN, Ganguly J. Studies on the relative biopotencies and intestinal absorption of different apo-beta-carotenoids in rats and chickens. Biochem J. 1976 Aug 15;158(2):377-83. doi: 10.1042/bj1580377. PMID 985434
- [Background] Arbuckle MR, McClain MT, Rubertone MV, Scofield RH, Dennis GJ, James JA, Harley JB. Development of autoantibodies before the clinical onset of systemic lupus erythematosus. N Engl J Med. 2003 Oct 16;349(16):1526-33. doi: 10.1056/NEJMoa021933. PMID 14561795
- [Background] Bjorklund H, Dalsgaard CJ, Jonsson CE, Hermansson A. Sensory and autonomic innervation of non-hairy and hairy human skin. An immunohistochemical study. Cell Tissue Res. 1986;243(1):51-7. doi: 10.1007/BF00221851. PMID 2417723
- [Derived] Imrich R, Alevizos I, Bebris L, Goldstein DS, Holmes CS, Illei GG, Nikolov NP. Predominant Glandular Cholinergic Dysautonomia in Patients With Primary Sjogren's Syndrome. Arthritis Rheumatol. 2015 May;67(5):1345-52. doi: 10.1002/art.39044. PMID 25622919